CLINICAL TRIAL: NCT05729763
Title: Three-dimensional Virtual Imaging to Improve the Accuracy of Standard CT-based Nephrometric Scores: a Prospective Multicentric Observational Study
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Francesco Porpiglia, Prof., San Luigi Gonzaga Hospital
Other Study IDs: 8193 02 06 - 07 Jun 2019
Record Dates: First submitted 2023-01-23; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Kidney Neoplasms; Carcinoma, Renal Cell
Keywords: minimally-invasive partial nephrectomy; nephrometry scores; 3D virtual imaging; HA3D; postoperative complications
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with localized renal tumor: Patients with localized renal tumor scheduled for minimally invasive partial nephrectomy in which 2D- and 3D-PADUA nephrometric score assessment was performed preoperatively
  Interventions: Other: 3D-PADUA nephrometric score; Other: 2D-PADUA nephrometric score

INTERVENTIONS:
Other: 3D-PADUA nephrometric score — Evaluation of the PADUA nephrometric score with 3D images
Other: 2D-PADUA nephrometric score — Evaluation of the PADUA nephrometric score with 2D images

SUMMARY:
STUDY DESIGN:

prospective multicentric observational

SAMPLE SIZE OF THE STUDY:

The estimated number of patients to enroll in the multicenter study is at least 270 patients (statistically calculated referring to the results of a monocentric analysis including 101 patients with the same design, already performed by the Coordinator Center).

NUMBER OF CENTERS INVOLVED:

Considering a total number of patients enrolled of at least 270, number of Centers to be involved: 5.

STUDY PROCEDURES:

3D virtual model rendering

* CT-scan images sent in DICOM format to MEDICS (Turin, Italy) after anonymization.
* Dedicated online platform available to upload the anonymized CT images, after registration.
* CT imaging processing by bioengineers and 3DVM building within 72 hours
* 3D-PDF download from the same online platform

Nephrometric score assessment

* All CT-scans and their 3DVMsevaluation in order to assess surgical complexity, as classified by the PADUA nephrometry score and its relative PADUA risk category.
* For each Center:

  * assessment of the PADUA score on the basis of the CT-scans (2D-NS) by one urologist;
  * assessment of the PADUA score on the basis of the 3DVMs (3D-NS) by another urologist.

Surgical intervention and pathological assessment

* Dedicated expert surgeon for each Center performing NSS to all patients with the same surgical technique.
* Dedicated uro-pathologist for each Center performing the histopathological evaluations of the specimens.

ELIGIBILITY:
Inclusion Criteria:

* four-phase (unenhanced, corticomedullary, nephrographic and urographic phases) contrast enhanced CT-scan

Exclusion Criteria:

* evidence of anatomical abnormalities, like horse-shoe shaped or ectopic kidney.
* preoperative imaging inadequate to perform a 3DVM (such as those with a CT-scan with >3 mm acquisition interval of the slices, or suboptimal difference of enhancement among the enhanced phases) or older than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized renal tumor scheduled for partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
PADUA nephrometry score calculated via 3D virtual modelling and standard bidimensional CT scan images | Baseline
  The PADUA nephrometry score predicts the risk of surgical and medical perioperative complications in patients who underwent partial nephrectomy.
  The PADUA nephrometry score evaluates different tumor characteristics:
  * Longitudinal (polar) location (Superior/inferior: 1pt; Middle: 2 pt),
  * Exophytic rate (>=50%: 1pt; <50%: 2pt; Endophytic: 3pt)
  * Renal rim (Lateral: 1pt; Medial: 2pt)
  * Renal sinus (Not involved: 1pt; Involved: 2pt)
  * Urinary collecting system (Not involved: 1pt; Dislocated/infiltrated: 2pt)
  * Tumor size (<=4 cm: 1pt; 4.1-7 cm: 2pt; >7: 3pt) The PADUA score, calculated as the sum of these parameters, stratify patients from PADUA 6 tumors, that have low risk of complications, to PADUA 14, with high risk of perioperative complications.

SECONDARY OUTCOMES:
To compare the occurrence of postoperative complications, assessed by Clavien-Dindo classification | 90 days after surgery
  The Clavien-Dindo classification evaluates severity of complications in 5 groups:
  * Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions;
  * Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications;
  * Grade III: Requiring surgical, endoscopic or radiological intervention (IIIa: Intervention not under general anesthesia; IIIb: Intervention under general anesthesia);
  * Grade IV Life-threatening complication requiring IC/ICU-management (IVa: single organ dysfunction; IVb: multiorgan dysfunction);
  * Grade V: Death of a patient.

CONTACTS AND LOCATIONS:
Locations (1):
- San Luigi Gonzaga Hospital, Orbassano, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided